CLINICAL TRIAL: NCT00457262
Title: Effects of Soy Protein on Serum paraoxonase1 Activity and Lipoproteins in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iran University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1344
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Last update posted 2007-04-06 (Estimated); Status verified 2007-03

CONDITIONS: Postmenopausal; Hyperlipidemia
Keywords: paraoxonase1 activity; LDL; HDL; postmenopausal women; postmenopausal women and hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: soy consumption

SUMMARY:
paraoxonase 1 is involved to prevent LDL and HDL oxidation,so increase of it's activity leads to lower risk of coronary heart disease.In postmenopausal women ,we have decrease of paraoxonase1 activity and soy proteins may increase paraoxonase1 activity

DETAILED DESCRIPTION:
In a double blind clinical randomised clinical trial with parallel design this study was done.52 postmenopausal women were randomly assigned to 50 g/d soy protein or placebo for 10 weeks.serum lipoproteins and pon1 activity were measured at baseline and 10th week.There were significant increase in PON! activity and significant decrease in LDL-C,LDL-C/HDL-C,TC/HDL-C and TG/HDL-C in soy group compare to placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Cessation of menes for more than 1 year, elevation for more than 1 year
* Elevation of FSH level
* Total cholesterol
* Triglyceride more than 200 mg/dl

Exclusion Criteria:

* Chronic disease (heart disease, cancer, diabetes, hepatic, kidney and thyroid disease)
* Antihypertensive drugs
* Antibiotics
* Lipid lowering drugs
* Sex hormone treatment
* Hysterectomy
* Diet rich in soy protein

Ages: 51 Years to 57 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42
Dates: Start 2006-01; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
decrease of LDL,increase of HDL,increase of paraoxonase 1

CONTACTS AND LOCATIONS:
Overall Officials: farzad Shidfar, Ph.D, Study Chair — assistant professor of nutrition,Iran university of medical sciences